CLINICAL TRIAL: NCT07397390
Title: A Prospective, Single-Arm Observational Study on the Effectiveness and Safety of the DKutting® LL Balloon in VEssel Preparation for CALcified Lesions in Infra-inguinal Arteries, the DkuLL CALVEP Study.
Brief Title: an Observational Study Evaluting the Effectiveness and Safety of DKutting LL Noval Scoring Balloon Angioplasty for Vessel Preparation Facilitated by IVUS on the Lower Limb Ischemia Patients With Calcified Lesions
Acronym: DkuLL CALVEP
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Ji Donghua, Medical Doctor, Chief Physician, The First Affiliated Hospital of Dalian Medical University, The First Affiliated Hospital of Dalian Medical University
Other Study IDs: PJ-KS-KY-2025-940(X); 20251012 (Other: The First Affiliated Hospital of Dalian Medical University)
Record Dates: First submitted 2026-01-29; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Femoral Artery Stenosis; Angioplasty; Cutting Balloon Angioplasty; Calcifications, Vascular; Intravascular Imaging Device; Peripheral Artery Disease; Infrapopliteal Arterial Occlusive Disease
Keywords: Peripheral Arterial Disease; Femoropopliteal Artery; Infrapopliteal Artery; Calcified Lesions; Scoring Balloon; Angioplasty; Vessel Preparation; Intravascular Ultrasound (IVUS); Observational Study
MeSH Terms: conditions — Vascular Calcification; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Dkutting LL treatment group: IVUS facilitated DKutting LL angioplasty
  Interventions: Device: DKutting LL scoring balloon angioplasty

INTERVENTIONS:
Device: DKutting LL scoring balloon angioplasty — Following the detection of calcified lesions by Intravascular Ultrasound (IVUS), and aided by its accurate measurements of lesion diameter and length, percutaneous transluminal angioplasty (PTA) was performed using the DKutting LL scoring balloon

SUMMARY:
This is a prospective, single-center, single-arm, observational study. It plans to enroll 58 patients with moderate to severely calcified lesions in the femoropopliteal or infrapopliteal arteries. Participants will be treated with the Scoring Balloon Dilatation Catheter manufactured by DK Medtech (Suzhou) Co., Ltd. The study aims to evaluate the immediate technical success rate and the improvement in lumen area and calcification burden as assessed by IVUS following percutaneous transluminal angioplasty with the scoring balloon. Clinical follow-ups will be conducted at discharge (or within 7 days), 1 month, 3 months, and 6 months post-procedure to observe secondary endpoints including the incidence of clinically driven target lesion revascularization and changes in Rutherford classification

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 85 years.
* Clinical diagnosis of lower extremity atherosclerotic arterial disease, with a Rutherford Classification of Category 2-5.
* The patient has provided written informed consent.
* Life expectancy > 1 year.
* Confirmed by clinical and CTA examination: de novo or restenotic lesions after PTA in the femoropopliteal or infrapopliteal arteries, with no stent implantation within 2 cm of the target lesion. Stenosis ≥70% or chronic total occlusion (CTO).
* Lesion confirmed by CTA and color Doppler to have moderate to severe calcification (PACSS Grade 3-4). Lesion can be single or tandem, with a total length ≤150 mm. Reference vessel diameter near the target lesion ≥2 mm.
* Allowable location of the target lesion: ≥1 cm distal to the common femoral artery bifurcation, and up to 10 cm above the ankle.
* If the lesion is below-the-knee (BTK), the inflow vessels must have no non-target lesions, or any non-target lesions must be successfully treated with the current device without vascular complications.
* No serious vascular complications such as flow-limiting dissection occur after pre-dilation of the target lesion.
* Presence of at least one reconstructible infrapopliteal runoff vessel patent to the ankle.

Exclusion Criteria:

* Allergy to contrast media.
* Coagulopathy; severe hepatic insufficiency (ALT or AST > 3 times the upper limit of normal).
* Cardiac insufficiency (New York Heart Association Class III-IV).
* Life expectancy < 1 year.
* Acute cardiovascular events (e.g., acute myocardial infarction, stroke) within the past 3 months; active gastrointestinal bleeding affecting the use of anticoagulant/antiplatelet therapy.
* Previous stent implantation or bypass surgery in the target vessel.
* Acute/subacute limb ischemia or thrombotic lesions.
* Contraindications to anticoagulation or antiplatelet therapy.
* Failure to cross the lesion with a guidewire during the procedure; anticipation that the IVUS catheter or DKutting balloon will be unable to cross the lesion after pre-dilation.
* Intraoperative occurrence of severe complications requiring conversion to other treatment methods (e.g., bypass surgery).
* Pregnant or lactating women.
* Active infection at the intended treatment site; foot wounds reaching WIfI Stage 3, or ankle/foot ulcers primarily of non-ischemic etiology.
* Patient withdrawal of informed consent.
* Planned amputation.
* Planned use of adjunctive therapy devices (e.g., atherectomy, laser).
* Participation in another interventional drug/device clinical study for lower limb arteries where the primary endpoint has not been reached, or planned participation in such a study.
* Patient is bedridden or unable to walk.
* Presence of an aneurysm in the ipsilateral limb vasculature.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lower limb ischemia caused by calcified lesion in femoral-popliteal and infra-popliteal artery
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2026-02-18 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
primary effectiveness outcome | immediately after the intervention
  Technical Success Rate:
  Definition: Immediate post-procedural residual stenosis ≤30% after dilation with the Scoring Balloon Dilatation Catheter or a conventional balloon catheter, and without the occurrence of severe flow-limiting dissection (Grade D-F according to the National Heart, Lung, and Blood Institute (NHLBI) classification).
primary safety outcome | 1 month
  Incidence of emergency target lesion revascularization, unplanned amputation above the ankle on the target side, or grade D or higher flow-limiting dissection or perforation requiring intervention

SECONDARY OUTCOMES:
Primary Patency Rate at 30 days | 1 month
  Freedom from clinically driven target lesion revascularization (CD-TLR) and a peak systolic velocity ratio (PSVR) of <2.4 on duplex ultrasound.
Primary Patency Rate at 6 months | 6 months
  Freedom from clinically driven target lesion revascularization (CD-TLR) and a peak systolic velocity ratio (PSVR) of <2.4 on duplex ultrasound.
Incidence of Clinically Driven Target Lesion Revascularization (CD-TLR) at 6 months | 6 months
  The need for repeat revascularization in patients with clinical symptoms, including recurrent rest pain, worsening ulcer, or new foot ulcer. Revascularization methods include endarterectomy, bypass surgery, or repeat endovascular angioplasty.
Change in Rutherford Classification at 1 month post-procedure | 1 month
  The proportion of patients showing an improvement of at least one category in the Rutherford Classification.
Intraoperative Complication Rate Related to Percutaneous Transluminal Angioplasty (PTA) | immediately after the intervention
  Includes the occurrence of immediate flow-limiting dissection (NHLBI Grade A-F) after dilation with the Scoring Balloon Catheter, vessel perforation caused by PTA, and distal embolism caused by PTA
ΔMLA (Change in Minimum Lumen Area) | immediately after the intervention
  Assessed by Intravascular Ultrasound (IVUS) to preliminarily evaluate the effectiveness of the DKutting balloon in vessel preparation for lower limb arterial calcified lesions, with the primary metric being the immediate post-procedural increase in MLA. Calculated as the difference in MLA measured by IVUS before and immediately after PTA.
ΔCalcification Burden Improvement | immediately after the intervention
  Assessed by IVUS, measured as the change in the arc of continuous calcification in the vessel wall cross-section. Calculated as the difference in the arc of continuous calcification (differentiating between intimal and medial) measured by IVUS before and immediately after PTA.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided